CLINICAL TRIAL: NCT05677568
Title: The CINCH-FMR Post-Market Registry: Percutaneous Repair in Functional Mitral Regurgitation
Acronym: CINCH-FMR
Status: Enrolling by invitation | Type: Observational
Sponsor: Cardiac Dimensions, Inc. (Industry)
Responsible Party: Sponsor
Organization: Cardiac Dimensions Pty Ltd (Industry)
Other Study IDs: PMS-1681-01
Record Dates: First submitted 2022-10-20; First posted 2023-01-10 (Actual); Last update posted 2023-03-14 (Actual); Status verified 2023-03

CONDITIONS: Functional Mitral Regurgitation; Mitral Regurgitation
Keywords: Functional Mitral Regurgitation; Mitral Regurgitation; Cardiac Dimensions; Carillon Mitral Contour System; CINCH; CINCH FMR; Carillon; CMCS
MeSH Terms: conditions — Mitral Valve Insufficiency

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

GROUPS / COHORTS (2):
- Prospective: "Prospective" patients are identified prior to undergoing the Carillon procedure and are only enrolled after being successfully implanted with the Carillon device (prior to hospital discharge). Prospective patients will have applicable medical history and details of the Carillon implant procedure collected from medical records. After the patient is discharged, the patient's primary care specialist (cardiologist) and clinical investigation site staff will coordinate follow-up evaluations. Patients will be evaluated at one (1), six (6), twelve (12) months per standard of care and with annual contact for an additional four (4) years, for a total of five (5) years to assess long-term safety of the Carillon implant.
  Interventions: Device: Carillon Mitral Contour System
- Retrospective/Prospective: "Retrospective/Prospective" patients are implanted with the Carillon device and are currently being followed-up per standard of care. These patients will have applicable data collected from their medical records, including medical history, data about the Carillon procedure and follow-up visit data done since receiving the Carillon implant. They will be evaluated prospectively per standard of care follow-up through five (5) years post-implant to assess long-term safety of the Carillon implant.
  Interventions: Device: Carillon Mitral Contour System

INTERVENTIONS:
Device: Carillon Mitral Contour System — The Cardiac Dimensions Carillon Mitral Contour System (CMCS) is a medical device and consists of the following components:
  1. A proprietary implant intended for permanent placement in the coronary sinus (CS)/great cardiac vein (GCV)
  2. A catheter-based delivery system which consists of a curved CMCS delivery catheter (3.2mm outer diameter) and a handle assembly
  3. A sizing catheter to enable the physician to estimate the overall CS/GCV dimensions so that an appropriately sized implant may be selected The implant is attached to the handle assembly and is delivered through the CMCS delivery catheter to the coronary vein along the posterolateral aspect of the mitral annulus. The implant is designed to re-shape the mitral annulus to reduce annular dilation and mitral regurgitation.
  Other Names: Cardiac Dimensions; CMCS

SUMMARY:
This is a retrospective and prospective, multi-center, post-market observational registry study. The primary objective of this post market registry is to continue to evaluate the long term safety and performance of the Carillon® Mitral Contour System® (CMCS) in a commercial (post market) setting.

DETAILED DESCRIPTION:
There are more than 22 million people worldwide with heart failure, including 5.3 million in the United States . Functional mitral regurgitation (MR), leakage of the mitral valve due to dilation of the left ventricle and annulus, occurs as a consequence of Heart Failure. Cardiac Dimensions has developed proprietary technology designed to address functional mitral regurgitation in a minimally invasive manner.

Previous studies have established that the Carillon® therapy has caused a significant reduction in functional MR. This reduction in MR results in clinically significant improvements in exercise tolerance, quality of life, and thus overall function in a symptomatic heart failure population.

To supplement the findings from these previous studies, Cardiac Dimensions is conducting this post-market registry of the Carillon® Mitral Contour System® (CMCS) in patients with functional mitral regurgitation. This registry is a retrospective and prospective, multi-center, clinical registry designed to further characterize the acute and long-term safety and performance profile of the CMCS. Up to 250 implanted patients will be enrolled at up to 40 centers located in the European Union and countries that recognize the CE-mark as a valid marketing authorization.

Patients enrolled in the registry have received the Carillon implant and will be assessed to document the long-term safety and performance of the device. These patients will be followed according to routine standard of care post procedure follow up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with functional mitral regurgitation (i.e., dilated cardiomyopathy), in accordance with CE-mark approved labeling
2. Patients implanted with the Carillon device
3. Patients must be ≥ 18 years old
4. Patients require informed consent prior to inclusion in this registry
5. Minimum baseline data, as described in CINCH Protocol, including:

   * Hemodynamic measures (by echocardiography)
   * Baseline must include the following measurements: MR grade, LVEF (%), LVEDD, LAD, and AP & ML diameters
   * NYHA Classification

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Up to 250 patients implanted with the Carillon implant.
Sampling Method: Non-Probability Sample
Enrollment: 250 (Estimated)
Dates: Start 2017-06-24 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2030-06-30 (Estimated)

PRIMARY OUTCOMES:
Death | 6 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 12 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 24 months
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 3 years
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 4 years
  All cause mortality including cardiovascular and non-cardiovascular death
Death | 5 years
  All cause mortality including cardiovascular and non-cardiovascular death
Serious adverse events | 6 months
  Number of procedure related or device related serious adverse events
Serious adverse events | 12 months
  Number of procedure related or device related serious adverse events
Change in New York Heart Association (NYHA) classification | 6, 12, and 24 months, and 3, 4, and 5 years
  Change in New York Heart Association (NYHA) Functional Classification at 6, 12, and 24 months, and 3, 4, and 5 years
Rate of Heart Failure Hospitalizations | 6 months
  Rate of hospitalization for heart failure
Rate of Heart Failure Hospitalizations | 12 months
  Rate of hospitalization for heart failure
Rate of Heart Failure Hospitalizations | 24 months
  Rate of hospitalization for heart failure
Rate of Heart Failure Hospitalizations | 3 years
  Rate of hospitalization for heart failure
Rate of Heart Failure Hospitalizations | 4 years
  Rate of hospitalization for heart failure
Rate of Heart Failure Hospitalizations | 5 years
  Rate of hospitalization for heart failure

SECONDARY OUTCOMES:
Change of MR Severity via Quantitative MR Variable: regurgitant volume (mL) | 6, 12, and 24 months, and 3, 4, and 5 years
  change in MR severity based in regurgitant volume as assessed by echocardiography in hospital, 6, 12, and 24 months, and 3, 4, and 5 years, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change of MR Severity via Quantitative MR Variable: regurgitant fraction (%) | 6, 12, and 24 months, and 3, 4, and 5 years
  change in MR severity based on regurgitant fraction (%) as assessed by echocardiography in hospital, 6, 12, and 24 months, and 3, 4, and 5 years, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change of MR Severity via Quantitative MR Variable: effective regurgitant orifice area (cm2 EROA) | 6, 12, and 24 months, and 3, 4, and 5 years
  change in MR severity based on effective regurgitant orifice area (cm2, EROA) as assessed by by Proximal Isovelocity Surface Area (PISA) via echocardiography in hospital, 6, 12, and 24 months, and 3, 4, and 5 years, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change of MR severity: Semi-Quantitative Parameter: Change in vena contract width | 6, 12, and 24 months, and 3, 4, and 5 years
  Change in vena contract width MR severity as assessed by echocardiography in hospital 6, 12, and 24 months, and 3, 4, and 5 years, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change of MR severity: Semi-Quantitative Parameter: Change in MV EVmax. | 6, 12, and 24 months, and 3, 4, and 5 years
  Change in MV EVmax MR severity as assessed by echocardiography in hospital, 6, 12, and 24 months, and 3, 4, and 5 years, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change of MR severity: Semi-Quantitative Parameter: Change in pulmonary vein flow. | 6, 12, and 24 months, and 3, 4, and 5 years
  Change in pulmonary vein flow MR severity as assessed by echocardiography in hospital, 6, 12, and 24 months, and 3, 4, and 5 years, in accordance with American Society of Echocardiography guidelines, compared to baseline.
Change in Left Atrial Area | 6, 12, and 24 months, and 3, 4, and 5 years
  Change in Left Atrial Area as assessed by echocardiography at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in Left Atrial Diameter | 6, 12, and 24 months, and 3, 4, and 5 years
  Change in Left Atrial Diameter as assessed by echocardiography at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in Left Atrial Volume Index | 6, 12, and 24 months, and 3, 4, and 5 years
  Change in Left Atrial Volume as assessed by echocardiography Index at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in Left Ventricular End Systolic Volume (LVESV) | 6,12, and 24 months, and 3, 4, and 5 years
  Change in Left Ventricular End Systolic Volume (LVESV) as assessed by echocardiography at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in Left Ventricular End Diastolic Volume (LVEDV) | 6,12, and 24 months, and 3, 4, and 5 years
  Change in Left Ventricular End Diastolic Volume (LVEDV) as assessed by echocardiography at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in Left Ventricular End Systolic Diameter (LVESD) | 6,12, and 24 months, and 3, 4, and 5 years
  Change in Left Ventricular End Systolic Diameter (LVESD) as assessed by echocardiography at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in Left Ventricular End Diastolic Diameter (LVEDD) | 6,12, and 24 months, and 3, 4, and 5 years
  Change in Left Ventricular End Diastolic Diameter (LVEDD) as assessed by echocardiography at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in Left Ventricular End Ejection Fraction (LVEF) | 6,12, and 24 months, and 3, 4, and 5 years
  Change in Left Ventricular End Ejection Fraction (LVEF) as assessed by echocardiography at 6, 12, and 24 months, and 3, 4, and 5 years over baseline
Change in exercise tolerance by walking | 6,12, and 24 months, and 3, 4, and 5 years
  Change in exercise tolerance as measured by meters walked in Six Minute Walk Test at 6,12, and 24 months, and 3, 4, and 5 years over baseline
Change in Quality-of-Life Overall Score | 6,12, and 24 months, and 3, 4, and 5 years
  Change in Quality of Life (QoL) score, as measured by Kansas City Cardiomyopathy Questionnaire (KCCQ) at 6,12, and 24 months, and 3, 4, and 5 years over baseline

CONTACTS AND LOCATIONS:
Overall Officials: Michael Haude, Prof. Dr., Principal Investigator — Rheinland Klinikum Neuss GmbH Lukaskrankenhaus
Locations (19):
- Germany (19):
  - Universitätsklinikum Aachen, Aachen
  - St. Marien Krankenhaus- Ahaus Vreden, Ahaus
  - Sana Klinikum Lichtenberg, Berlin
  - Klinikum Links der Weser, Bremen
  - Kardiovaskular Zentrum Darmstadt, Darmstadt
  - Herzzentrum Dresden, Dresden
  - Cardiovascular Center Frankfurt, Frankfurt
  - Universtitätsklinikum Frankfurt, Frankfurt
  - Hostpital zum Heiligen Geist, Fritzlar
  - Asklepios Klinik Altona, Hamburg
  - Kath. Marienkrankenhaus GmbH- Hamburg, Hamburg
  - Krankenhaus Agatharied GmbH, Hausham
  - Universitätsklinikum Schleswig-Holstein, Campus Kiel, Kiel
  - Universitätsklinikum Leipzig, Leipzig
  - Universitätsmedizin Mainz, Mainz
  - Universitätsmedizin Mannheim, Mannheim
  - Rheinland Klinikum Neuss GmbH- Lukaskrankenhaus, Neuss
  - Universitätsklinikum Ulm, Ulm
  - Josefs Hospital Wiesbaden, Wiesbaden

IPD SHARING:
Plan to Share IPD: No
No plans for sharing